CLINICAL TRIAL: NCT05947929
Title: Aerobic Exercise Verus Acupuncture on the Quality of Life in Women Suffering From Irritable Bowel Syndrome [NCT ID Not Yet Assigned]
Brief Title: Aerobic Exercise Verus Acupuncture on the Quality of Life in Women Suffering From Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, manal nasser husain, Principal Investigator, Cairo University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IBS
Record Dates: First submitted 2023-07-08; First posted 2023-07-17 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: Acupuncture; Aerobic exercise; Quality of life
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treadmill exercise Group (Experimental): 30 women will perform treadmill exercise following low food map diet three times \weak for 3 months
  Interventions: Other: Aerobic excise
- acupuncture Group (Experimental): 30 women will receive acupuncture session following low food map diet three times \ weak for 3 months.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: Aerobic excise — the treadmill exercises three times a week for 12 weeks) based on the Following protocol: Intensity exercise: determined by karvonen formula: Exercise heart rate = [(A-B) × desired intensity] + B [A represents maximum heart rate (220-age) and B for resting heart rate (average of three measurements)]. The desired intensity will be at 50- 70%. Heart rate was measured by pulse-meter to detect pulse rate before exercise (Resting HR)].
  Arms: treadmill exercise Group
Other: acupuncture — the acupuncture needles will be inserted through the adhesive pads. The acupuncture needles used in the study are 40 mm in length and 0.30 mm in diameter and manufactured by Suzhou Hwato Medical Instruments Co. Ltd (Suzhou, China). The following acupoints will be used: DU20 (Baihui), ST36 (Zusanli), ST37 (Shangjuxu), SP6 (Sanyinjiao), ST25 (Tianshu), and LR3 (Taichong).
  Arms: acupuncture Group

SUMMARY:
To compare the effect of aerobic exercise and the acupuncture on the quality of life in women with irritable bowel syndrome

DETAILED DESCRIPTION:
Patients with IBS have a higher prevalence of migraine, fibromyalgia and depression.

Donald et al. have shown that physically active elderly participants were less likely to be constipated than their less active counterparts.

On the quality of life Physical activity has also been shown to reduce mouth-to-anus transit time and among individuals with constipation, higher levels of physical activity were found to be associated with improved physical functioning and health perceptions. Similarly, other finding studies are not consistent with some small observational studies which have failed to report positive associations between exercise and constipation, reported that orocecal transit time was accelerated during mild exercise. Of some relevance to the findings reported here is a recent randomized controlled trials (RCT) that found walking to be an effective intervention for improving the degree of bowel cleansing in preparation for a colonoscopy. There is a contradiction between studies.

However, study results on acupuncture in IBS are mixed, and more larger trials are needed to fully support the claims of acupuncture in helping with IBS there's a contradiction between the studies so, the present study will be conducted to compare the effect of aerobic exercise and acupuncture on women with irritable bowel syndrome and to solve the contradiction. .

ELIGIBILITY:
Inclusion Criteria:1- Sixcity Females with mild and moderate IBS from Owsim General Hospital. Being able to increase the level of physical activity.

2- Their age will be 35 to45 years old 3- Stable vital signs ( blood pressure , respiratory rate and temperature) 4- BMI <30 (Fani et al., 2019) 5- Patients meeting the Rome III diagnostic criteria for IBS. 6- Baseline IBS-SSS score from 75to 299(mild and moderate) 7- No medication for IBS (except for emergency) within at least 2 weeks ago. 8- No acupuncture therapy within 3 months prior to study recruitment (Lixia et al., 2018).

9- NO following any type of diet within 3 months prior to the treatment

-

Exclusion Criteria: Patients meeting any of the following criteria will be excluded

1. The patient has a history of rheumatic diseases in the lower limb.
2. Having a history of metabolic, neurologic, cardiovascular, respiratory, renal, and lung problems which would prevent them from participating in aerobic exercises.
3. Having a history of knee injury or knee surgery during the past year or having a history of joint replacement in any of the joints of the lower limb.
4. Having a history of fracture in the lower limb during the past six months
5. Major vision disorders.
6. Hereditary or acquired musculoskeletal disorders in the lower limb.
7. Organic gastrointestinal disorders.
8. Using drugs that would affect metabolism or balance.
9. Using assistive devices for walking (Fani et al., 2019)
10. Intestinal organic diseases or systemic diseases affecting gastrointestinal motility (such as gallbladder pancreatitis, hyperthyroidism, diabetes, chronic renal insufficiency, and nervous system diseases).
11. History of abdominal or rectal anus surgery.
12. pregnancy or breastfeeding, and post-partum 12 months,
13. Installation of the cardiac pacemaker.
14. metal allergy, and fear of the needle.

    -

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 30 female patients with IBS
Enrollment: 60 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Assessing the change in pain intensity | at baseline and after 3 months of intervention
  By using visual anaglouge scale. The visual analog scale (VAS) is the VAS, which consists of a line, usually 10 cm long, ranging from no pain or discomfort (zero) , to the worst pain that could possibly feel (10)
Assessing the change in level of exertion during physical activity | at baseline and after 3 months of intervention
  The Borg scale is a numerical scale that ranges from 6 to 20 where 6 means "no exertion at all" and 20 means "maximal exertion." When a measurement is taken, a number is chosen from the following scale by an individual that best describes their level of exertion during physical activity.
Assessing the change in Irritable Bowel Syndrome Symptom Severity | at baseline and after 3 months of intervention
  by Irritable Bowel Syndrome Symptom Severity Score (IBS- SSS). Patients completed IBS-SSS questionnaire for assessing their eligibility for the study. IBS-SSS questionnaire contains five questions which would measure pain severity, pain frequency, abdominal bloating, bowel habit dissatisfaction, and life interference using Visual Analogue Scale (VAS). The mean score of each item ranges from 0 to 100 and the total mean score of the questionnaire ranges from 0 to 500; higher scores indicates more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Manal Nasser Hussein, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic faculty of physical therapy cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided